CLINICAL TRIAL: NCT05134987
Title: A Multiple Dose Study Investigating Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0363-0845 in Participants With Type 1 Diabetes
Brief Title: A Multiple Dose Study Investigating Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0363-0845 in Participants With Type 1 Diabetes Pharmacokinetics and Pharmacodynamics: How Insulin NNC0363-0845 is Transported Throughout the Body and How It Works
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1845-4886; U1111-1266-4162 (Other: World Health Organization (WHO)); 2021-003271-33 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0363-0845 followed by insulin detemir (Experimental): Participants will get subcutaneous (under the skin) injections of insulin NNC0363-0845 (study medicine) up to 6 times daily for 3 days. After a 4-21 days wash-out period with no injections they will get subcutaneous injections of insulin detemir up to 6 times daily for 3 days.
  Interventions: Drug: NNC0363-0845
- Insulin detemir followed by NNC0363-0845 (Experimental): Participants will get subcutaneous (under the skin) injections of insulin detemir up to 6 times daily for 3 days. After a 4-21 days wash-out period with no injections they will get subcutaneous injections of NNC0363-0845 (study medicine) up to 6 times daily for 3 days.
  Interventions: Drug: Insulin detemir

INTERVENTIONS:
Drug: NNC0363-0845 — Participants will receive 0.5 nmol/kg NNC0363-0845 s.c. (subcutaneous - under the skin) every 4 hours up to 6 times daily (i.e. 3 nmol/kg/day) for 3 days The study will last for about 6 weeks up to a maximum of 14 weeks
  Arms: NNC0363-0845 followed by insulin detemir
Drug: Insulin detemir — Participants will receive 0.083 U/kg insulin detemir s.c. (subcutaneous - under the skin) every 4 hours up to 6 times daily (i.e. 0.5 U/kg/day) for 3 days The study will last for about 6 weeks up to a maximum of 14 weeks
  Arms: Insulin detemir followed by NNC0363-0845

SUMMARY:
This study is designed to investigate the movement of insulin NNC0363-0845 throughout the body and how it works for the treatment of type 1 diabetes mellitus.

The aim of the study is to improve clinical outcomes for patients with type 1 diabetes mellitus by better controlling the blood sugar levels.

Participants will get insulin NNC0363-0845 as well as insulin detemir (Levemir®). NNC0363-0845 is a new insulin molecule designed to provide blood sugar-dependent insulin action, while insulin detemir is commonly used and prescribed by doctors.

Participants will get subcutaneous (under your skin) injections of insulin NNC0363-0845 (study medicine) up to 6 times daily for 3 days, and of insulin detemir up to 6 times daily for another 3 days. Which medication participants receive first and which second, insulin NNC0363-0845 or insulin detemir, is decided by chance.

The study will last for about 6 weeks up to a maximum of 14 weeks. Participants will have 2 in-house visits (where participants will stay at the site for 4 nights) and 5 outpatient visits with the study doctor. Participants will have frequent contact with the study doctor during the study.

During the in-house visits, two intravenous catheters (a thin tube inserted into a vein) will be inserted for blood sampling and infusions.

Interested parties may not participate in the study if the study doctor believes it will affect their health negatively.

Women cannot take part if they are of childbearing potential.

ELIGIBILITY:
Key inclusion criteria:

* Male participant or female participant of non-childbearing potential. Non-child-bearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 1 diabetes mellitus 1 year or more before screening.
* Current daily basal insulin treatment greater than 0.2 and below or equal to 0.5 (I)U/kg/day.
* Current total daily insulin treatment between 0.4 and 0.8 (I)U/kg/day (both inclusive).
* Body mass index between 18.5-29.9 kg/m^2 (both inclusive).
* HbA1c (glycated haemoglobin) below or equal to 8.0%.

Key exclusion criteria:

* Male of reproductive age who, or whose female partner(s), is not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice). Adequate contraceptive measures include that the male participant uses a condom during intercourse and that the partner practices adequate contraception (risk of pregnancy must be lower than 1%). In addition, participants must not donate sperm for the duration of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
AUCPG,0.5-2h Area under the plasma glucose-time curve at steady concentrations | From 0.5 to 2 hours after initiation of meal glucose appearance test (visit 4 day 3 and visit 5 day 3)
  messured in h*mmol/L

SECONDARY OUTCOMES:
AUCPG,0-1h Area under the plasma glucose-time curve at steady concentrations | From 0 to 1 hour after initiation of meal glucose appearance test (visit 4 day 3 and visit 5 day 3)
  messured in h*mmol/L
AUCPG,0-2hArea under the plasma glucose-time curve at steady concentrations | From 0 to 2 hours after initiation of meal glucose appearance test (visit 4 day 3 and visit 5 day 3)
  messured in h*mmol/L
AUCPG,0-4h Area under the plasma glucose-time curve at steady concentrations | From 0 to 4 hours after initiation of meal glucose appearance test (visit 4 day 3 and visit 5 day 3)
  messured in h*mmol/L
∆PGav,0-1h Mean change in plasma glucose at steady concentrations | From 0 to 1 hour after initiation of meal glucose appearance test (visit 4 day 3 and visit 5 day 3)
  messured in mmol/L
∆PGav,0-2h Mean change in plasma glucose at steady concentrations | From 0 to 2 hours after initiation of meal glucose appearance test (visit 4 day 3 and visit 5 day 3)
  messured in mmol/L
Number of adverse events | From first IMP administration until 16 hours after last IMP administration (visit 4 day 3 and visit 5 day 3)
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com